CLINICAL TRIAL: NCT06909968
Title: Identification of Palliative Care Needs and Prognostic Factors of Survival in Tailoring Appropriate Interventions in Advanced Oncological, Renal and Pulmonary Diseases
Status: Completed | Type: Observational
Sponsor: Istituto Romagnolo per lo Studio dei Tumori Dino Amadori IRST S.r.l. IRCCS (Other)
Responsible Party: Sponsor
Other Study IDs: IRST100.45
Record Dates: First submitted 2025-03-20; First posted 2025-04-04 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-10

CONDITIONS: Cancer; Chronic Renal Failure; Chronic Obstructive Pulmonary Disease; Idiopathic Pulmonary Fibrosis
Keywords: palliative care; appropriateness; cancer; chronic pulmonary failure; chronic renal failure
MeSH Terms: conditions — Neoplasms; Kidney Failure, Chronic; Pulmonary Disease, Chronic Obstructive; Idiopathic Pulmonary Fibrosis | interventions — Palliative Care

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Cancer patients: cancer patients with first diagnosis of inoperable locally advanced and/or metastatic non-small cell lung cancer, or gastric cancer or pancreatic adenocarcinoma
  Interventions: Other: palliative care
- Chronic pulmonary failure: patients with advanced chronic respiratory failure, caused by chronic obstructive pulmonary disease (COPD) or idiopathic pulmonary fibrosis (IPF).
  Interventions: Other: palliative care
- Chronic renal failure: patients with advanced chronic renal failure
  Interventions: Other: palliative care

INTERVENTIONS:
Other: palliative care — As this study is intended to be observational (not interventional), the patient's medical record will be the source of all data to be recorded.
  No additional procedures/patient visits should be planned in the study with respect to clinical practice.
  Two tools will be used to to analyze appropriateness and timeliness of progressive palliative care approach: NECPAL CCOMS-ICO(©), specific for the assessment of needs in palliative care, and the PaP score, for the assessment of prognosis.

SUMMARY:
This is a prospective observational study done on 3 patient populations (cancer, chronic pulmonary and renal disease). All patients will be treated and monitored according to the local clinical practice. No additional procedures/patient visits in comparison with the usual clinical practice are planned for the study.

DETAILED DESCRIPTION:
This is a prospective observational study done on 3 patient populations (cancer, chronic pulmonary and renal disease). All patients will be treated and monitored according to the local clinical practice. No additional procedures/patient visits in comparison with the usual clinical practice are planned for the study. The primary objective is to analyze appropriateness and timeliness of progressive palliative care approach (initially simultaneously with ongoing disease-oriented treatment and subsequently possibly as the only modality of care to avoid aggressiveness of care) in patients with:

* First diagnosis of advanced metastatic non-small cell lung cancer, or advanced gastric cancer or advanced pancreatic adenocarcinoma
* advanced chronic respiratory failure, caused by chronic obstructive pulmonary disease (COPD) or idiopathic pulmonary fibrosis (IPF).
* advanced chronic renal failure

ELIGIBILITY:
Inclusion Criteria:

* Both sex;
* All ethnic background;
* Age ≥18 years;
* Subjects who are, in the opinion of the Investigator, able to understand this study and to cooperate with the study procedures;
* Written informed consent;
* Not receiving care from the palliative care service

Inclusion Criteria specific for POPULATION A:

* Diagnosis of inoperable locally advanced and/or metastatic non-small cell lung cancer, or gastric cancer or pancreatic adenocarcinoma within the previous eight weeks, any T, any N, M+ or T4 inoperable (neoadjuvant excluded);
* Life expectancy >2 months;

Inclusion Criteria specific for POPULATION B:

* Diagnosis of chronic obstructive pulmonary disease (COPD) with at least two of these characteristics: age > 70 years, FEV1 <30 % predicted, oxygen-therapy dependency, > 1 admission/year in hospital for COPD exacerbated, congestive heart failure and/or other comorbidity, weight loss/cachexia, reduced functional autonomy, increase dependence.
* or idiopathic pulmonary fibrosis (IPF) diagnosis with at least two of these characteristics: age > 70 years, histological pattern "UIP" (if known), dependence on oxygen-therapy, radiological aspect of "Honeycomb" to the HRTC of the thorax, reduced functional autonomy, increased dependence.

Inclusion Criteria specific for POPULATION C:

- Diagnosis advanced chronic renal failure with at least two of these characteristics: age > 75 years, advanced malignancy, severe malnutrition, cardiac or pulmonary pathology terminal, Multiple Organ Failure in Intensive Care.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: * Population A: cancer patients with first diagnosis of inoperable locally advanced and/or metastatic non-small cell lung cancer, or gastric cancer or pancreatic adenocarcinoma.
  * Population B: patients with advanced chronic respiratory failure, caused by chronic obstructive pulmonary disease (COPD) or idiopathic pulmonary fibrosis (IPF).
  * Population C: patients with advanced chronic renal failure.
Sampling Method: Non-Probability Sample
Enrollment: 178 (Actual)
Dates: Start 2020-12-14 (Actual); Primary Completion 2025-02-26 (Actual); Study Completion 2025-10-17 (Actual)

PRIMARY OUTCOMES:
Evaluating PaP (Palliative Prognostic) and NECPAL CCOMS-ICO(©) scores to analyze the appropriateness of progressive palliative care approach | 55 months
  Initially simultaneously with ongoing disease-oriented treatment and subsequently as the only modality of care to avoid aggressiveness of care.
Evaluating PaP (Palliative Prognostic) and NECPAL CCOMS-ICO(©) scores to analyze timeliness of progressive palliative care approach | 55 months
  Initially simultaneously with ongoing disease-oriented treatment and subsequently as the only modality of care to avoid aggressiveness of care.

CONTACTS AND LOCATIONS:
Overall Officials: Marco C Maltoni, MD, Study Chair — IRST IRCCS
Locations (5):
- Italy (5):
  - Rete Cure Palliative AUSL Bologna, Bologna, BO
  - U.O. Nefrologia, Dialisi e Trapianto Renale, Policlinico Sant'Orsola, Bologna, BO
  - U.O. Pneumologia e Terapia Intensiva Respiratoria, Policlinico Sant'Orsola, Bologna, BO
  - U.O. Nefrologia e Dialisi, Ospedale Morgagni-Pierantoni - Ospedale M. Bufalini, Forlì, FC
  - IRST IRCCS UO Cure Palliative, Meldola